CLINICAL TRIAL: NCT03509753
Title: Prebiotic Fiber to Prevent Pathogen Colonization in the Intensive Care Unit (ICU)
Brief Title: Prebiotic Fiber to Prevent Pathogen Colonization in the ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Daniel Freedberg, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAR5162; 1K23DK111847-01 (NIH)
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Sepsis
Keywords: Prebiotic fiber
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Fiber (Experimental): Per 10 ounces of feed: 4 g oat-soy fiber with 45% short-chain fructooligosaccharides, 296 kCal, 19 g protein, 8 g fat, and 39 g carbohydrates. Feed rate/duration individualized for each patient.
  Interventions: Dietary Supplement: High Fiber
- Low Fiber (Active Comparator): Per 10 ounces of feed: 0 g fiber, 296 kCal, 19 g protein, 8 g fat, and 39 g carbohydrates. Feed rate/duration individualized for each patient.
  Interventions: Dietary Supplement: Low Fiber

INTERVENTIONS:
Dietary Supplement: High Fiber — See intervention description.
  Arms: High Fiber
Dietary Supplement: Low Fiber — See intervention description.
  Arms: Low Fiber

SUMMARY:
This is a pilot trial testing enteral feeds that are high versus low in prebiotic fiber in 20 critically ill adults. The long-term goal is to determine the efficacy of fiber for the prevention of pathogen colonization/infection in the ICU.

DETAILED DESCRIPTION:
This study will test prebiotic fiber in 20 adults who are receiving broad-spectrum antibiotics in the medical or surgical ICU by open-label randomization of patients to approximately 20 g prebiotic fiber/day including 45% short-chain fructooligosaccharides versus 0 g fiber/day by providing one of two feeds. Per 10 ounces of feed, both the high and low fiber feeds contain identical micronutrients and have 296 kilocalorie (kCal), 19 g protein, 8 g fat, and 39 g carbohydrates. The sole difference is that the fiber-containing feed has 4 g fiber including 45% short-chain fructooligosaccharides per 10 ounces whereas the other feed has 0 g fiber. Randomization will take place at the time the order for enteral feeding is placed. Rather than supplying the feed itself, the investigators will supply a randomized recommendation for a feed type (i.e., high vs low fiber) and the feed will be obtained from the hospital pharmacy in the usual manner. Determination of the feed rate and duration will be decided on the individual patient's needs by the treating ICU team. The primary outcome will be to determine whether high fiber feeds alter the gut microbiome in the face of antibiotics and critical illness, calculated by comparing within-individual microbiome differences from baseline to Day 3 in each intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Medical or surgical ICU patients ≥18 years old at our institution;
* Receiving broad-spectrum antibiotics at the time of enrollment;
* Deemed appropriate for the study by the treating ICU team;
* With capacity to give consent or have an appropriate surrogate;
* Able to undergo assessment within 4 hours of the order for enteral feeds;
* Expected to receive enteral feeds for ≥3 days but not yet receiving them.

Exclusion Criteria:

* Inability to receive enteral feeds;
* Celiac disease or known allergy to fiber;
* Surgery involving the intestinal lumen within 30 days;
* Limited treatment goals (i.e., do-not-resuscitate (DNR), do-not-intubate (DNI), or no escalation of care);
* Lack of capacity to consent and lack of an appropriate legally authorized representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change in microbiome measured by LEfSe | Baseline and Day 3
  An untargeted hierarchical linear discriminant analysis effect size algorithm (LEfSe) will be used to test for within-individual taxonomic differences comparing baseline to Day 3 in the high fiber group as it is an established method for identifying differences in bacterial taxa between any two groups. For those taxa which are significantly altered on LEfSe, the relative change in the high fiber group versus the relative change in the low fiber group will be computed using a rank-sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E. Freedberg, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Sequencing data and corresponding metadata will be made available through the Short Read Archive (SRA) section of the National Center for Biotechnology Information (NCBI) at the time of publication of the study results.
Time Frame: Data will be made available at the time of publication.
Access Criteria: Open.